CLINICAL TRIAL: NCT04121715
Title: A Prospective, Multicenter, Randomized Controlled Trial of Fastigial Nucleus Stimulation in Patients With Coronary Heart Disease
Brief Title: Fastigial Nucleus Stimulation for Coronary Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Collaborators: the Third Hospital of Mianyang (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ScHFPC-16PJ176
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Coronary Disease
Keywords: coronary heart disease; fastigial nucleus stimulation; inflammatory factors
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard medication (Active Comparator): standard medication:Refer to the "Guidelines for Rational Use of Coronary Heart Diseases"
  Interventions: Drug: Standard treatment
- standard medication+fastigial nucleus stimulation (Experimental): 1. fastigial nucleus stimulation:Use fastigial nucleus stimulation therapy device (Shanghai Renhe Medical Equipment Co., Ltd. CVFT series), each stimulation for 30 min, once a day, each patient treatment for about 20 days.
  2. standard medication:Refer to the "Guidelines for Rational Use of Coronary Heart Diseases"
  Interventions: Device: Fastigial Nucleus Stimulation; Drug: Standard treatment

INTERVENTIONS:
Device: Fastigial Nucleus Stimulation — Select mode 3, frequency 136, intensity below 90, ratio 1.0-2.0, based on the patient's no discomfort. The main pole is attached to the bilateral mastoid, and the auxiliary pole is attached to the bilateral internal cave. Non-invasive introduction of bio-electricity into the cerebellar nucleus for stimulation
  Other Names: Standard treatment
  Arms: standard medication+fastigial nucleus stimulation
Drug: Standard treatment — Refer to the "Guidelines for Rational Use of Coronary Heart Diseases".rational selection of antiplatelet drugs, statins, etc. according to the patient's condition

SUMMARY:
To observe the effects of fastigial nucleus stimulation on serum inflammation, oxidative stress related factors, cardiac autonomic function and prognosis in patients with coronary heart disease

DETAILED DESCRIPTION:
In recent years, with the improvement of the material living standards of the investigators residents and the change of working lifestyle, the prevalence and mortality of coronary heart disease (CHD) in urban and rural residents in China have increased year by year. According to statistics, the number of patients with coronary heart disease in China is currently 11 million. Coronary heart disease has become a major health problem in China. At present, it is found that inflammatory reaction and oxidative stress factors are involved in the occurrence and development of coronary heart disease, and their indicators such as heart rate variability are related to the prognosis of coronary heart disease. Fastigial nucleus stimulation (FNS) has been widely used in the treatment of various diseases such as cerebrovascular disease, migraine, and eye diseases. The study found that FNS can reduce inflammatory cytokines and oxidative stress factors in ischemic myocardium and improve heart rate variability in rats with myocardial infarction. The aim of this study was to investigate whether FNS can improve the aforementioned indicators and clinical outcomes in patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography was performed after admission, and coronary heart disease was diagnosed (coronary angiography showed at least one coronary artery with a diameter reduction of ≥50% from more than two different angles)
* Patients and their families agreed and signed informed consent

Exclusion Criteria:

* Severe chronic heart failure, and LVEF <30%
* Body temperature > 38 ° C and / or combined with severe infection in any system
* Severe liver and kidney dysfunction
* Malignant tumor
* Autoimmune diseases
* High blood pressure and diabetes with severe comorbidities
* Use of implantable electronic devices
* Intracranial implanted vascular stents
* Surface treatment electrode conductive materials Allergic or mastoid skin lesions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Observe the changes of serum IL-6 after treatment. | baseline,1month
  Observe the changes of serum IL-6 levels（pg/ml）after treatment in the two groups of patients.
Observe the changes of serum hs-CRP after treatment. | baseline,1month
  Observe the changes of serum hs-CRP levels（mg/l）after treatment in the two groups of patients.
Observe the changes of serum TNF-α after treatment. | baseline,1month
  Observe the changes of serum TNF-α levels（pg/ml）after treatment in the two groups of patients.
Observe the changes of serum Lp-PLA2 after treatment. | baseline,1month
  Observe the changes of serum Lp-PLA2 levels（ng/ml）after treatment in the two groups of patients.
Observe the changes of serum SOD（Superoxide dismutase） after treatment. | baseline,1month
  Observe the changes of serum SOD levels（ng/ml）after treatment in the two groups of patients.
Observe the changes of serum GPX（Glutathione peroxidase） after treatment. | baseline,1month
  Observe the changes of serum GPX levels（ng/ml）after treatment in the two groups of patients.
Observe the changes of serum MDA（Malondialdehyde） after treatment. | baseline,1month
  Observe the changes of serum MDA levels（nmol/ml）after treatment in the two groups of patients.
Observe the changes of serum AOPP（Advanced oxidation protein product） after treatment. | baseline,1month
  Observe the changes of serum AOPP levels（umol/l）after treatment in the two groups of patients.
Observe the changes of SDNN（Standard Deviation of the NN intervals） after treatment. | baseline,1month
  Observe the changes of SDNN（ms）after treatment in the two groups of patients.
Observe the changes of SDANN（Standard Deviation of mean NN intervals in 5-minute recordings） after treatment. | baseline,1month
  Observe the changes of SDANN（ms）after treatment in the two groups of patients.
Observe the changes of SDNN In（Average of the standard deviation of the NN interval every 5 minutes） after treatment. | baseline,1month
  Observe the changes of SDNN In（ms）after treatment in the two groups of patients.
Observe the changes of rMSSD（square root of the mean squared differences of successive NN intervals） after treatment. | baseline,1month
  Observe the changes of rMSSD（ms）after treatment in the two groups of patients.
Observe the changes of pNN50（Percentage of the difference between adjacent RR intervals >50ms ） after treatment. | baseline,1month
  Observe the changes of pNN50（%）after treatment in the two groups of patients.

SECONDARY OUTCOMES:
Follow-up rate of major cardiovascular events | 12months
  The improvement of symptoms and the in-stent restenosis, myocardial infarction, readmission due to heart failure, and mortality were observed in the two groups after 12 months of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Runfeng Zhang, Ph.D, Study Chair — the Third Hospital of Mianyang; Wensong Li, master, Principal Investigator — the Third Hospital of Mianyang; Xin Lei, master, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College; Xiaoju Liu, master, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College
Locations (1):
- The Third Hospital of Mianyang, Mianyang, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6months of study completion
Access Criteria: Data access requests will be reviewed by an external independent Reviwe Panel.Requestors will be required to sign a Data Access Agreement
URL: http://bethesda.org